CLINICAL TRIAL: NCT00838214
Title: Efficacy and Safety of Budesonide Capsules (3x3mg/d)Versus Prednisone in Patients With a Diagnose of Active Autoimmune Hepatitis. A Double-blind, Randomized, Active-controlled, Multicentre Study
Brief Title: Budesonide 3x3mg/d Versus Prednisone in Active Autoimmune Hepatitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Markus Proels, Dr. Falk Pharma, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUC-38/AIH
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Autoimmune Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune | interventions — Budesonide; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- budesonide (Experimental): 3mg capsules 3x/day for 6 months
  Interventions: Drug: budesonide
- prednisone (Active Comparator): 5mg tablet, 40mg starting dose titrated to 10mg over 3 months
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: budesonide — 3mg capsule, 3x per day for 6 months
  Arms: budesonide
Drug: prednisone — 5mg tablet, 40mg starting dose per day, titration to 10mg per day within 3 months
  Arms: prednisone

SUMMARY:
This is a multicentre, multinational clinical study. It comprised two consecutive segments (A and B). Segment A was designed as a randomized, double-blind, double-dummy, active-controlled, two-arm parallel-group study. The patients received either budesonide or prednisone for 6 months. During segment B all patients received budesonide as an open treatment for additional 6 months.

In this confirmatory study the proportion of patients with complete response was compared between the two treatment groups. Complete response was defined as biochemical remission (=serum levels of ASAT and ALAT within normal ranges) at the individual last visit of segment A and lack of steroid specific side effects throughout segment A.

ELIGIBILITY:
Inclusion Criteria:

* age 10 to 70 years
* Diagnosis of acute AIH according to Alvarez score
* normal range of TPMT activity
* normal ACTH test
* negative pregnancy test at screening for females of childbearing potential
* written informed consent

Exclusion Criteria:

* presence of Hepatitis A, B, C, E or G virus infection
* liver cirrhosis or clinical signs of portal hypertension
* PBC
* PSC
* history of hypersensitivity to the study medication

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2001-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Biochemical remission (=serum levels of ASAT and ALAT within normal ranges) at the individual last visit of Segment A and lack of steroid specific side effects | 6 months

SECONDARY OUTCOMES:
incidence of biochemical remission | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Manns, Professor, Principal Investigator — University Hospital
Locations (1):
- Medical School Hannover, Hanover, Lower Saxony, Germany

REFERENCES:
- [Result] Manns MP, Woynarowski M, Kreisel W, Lurie Y, Rust C, Zuckerman E, Bahr MJ, Gunther R, Hultcrantz RW, Spengler U, Lohse AW, Szalay F, Farkkila M, Prols M, Strassburg CP; European AIH-BUC-Study Group. Budesonide induces remission more effectively than prednisone in a controlled trial of patients with autoimmune hepatitis. Gastroenterology. 2010 Oct;139(4):1198-206. doi: 10.1053/j.gastro.2010.06.046. Epub 2010 Jun 22. PMID 20600032
- [Derived] Woynarowski M, Nemeth A, Baruch Y, Koletzko S, Melter M, Rodeck B, Strassburg CP, Prols M, Wozniak M, Manns MP; European Autoimmune Hepatitis-Budesonide Study Group. Budesonide versus prednisone with azathioprine for the treatment of autoimmune hepatitis in children and adolescents. J Pediatr. 2013 Nov;163(5):1347-53.e1. doi: 10.1016/j.jpeds.2013.05.042. Epub 2013 Jun 28. PMID 23810723